#### STATISTICAL ANALYSIS PLAN

# A DOSE-FINDING STUDY FOR LEVODOPA, CARBIDOPA AND **ODM-104** TEST FORMULATIONS AFTER REPEATED ADMINISTRATION IN HEALTHY MALES

| 3112005 |
|----------|
| COMDOS 1 |

Phase I study

Standard: GCP

The statistical analysis plan is approved and valid from the date of the last esignature on the last page

Clinical Study Director: Aila Holopainen
Study Statistician: Mikko Vahteristo
Development Leader: Juha Ellmén

Statistical analysis plan written by: Mikko Vahteristo

Property of Orion Corporation Sponsor: ORION PHARMA

#### Confidential

This documentation and other submissions made to you by Orion Corporation contain confidential information which Orion Corporation considers trade secrets and exclusive property of Orion Corporation or its principals and which may not be disclosed to third parties nor used for purposes other than that for which it has been submitted, without the express prior written consent of Orion Corporation, unless specifically provided for otherwise by law.

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 1/28

# **Table of contents**

| 1 | Abbreviations | 4 |
|---|---|---|
| 2 | General remarks | 4 |
| 3 | Overall study design and plan | 4 |
| 4 | Study objectives | 5 |
| 4.1 | Primary objective | 5 |
| 4.2 | Secondary objectives | 5 |
| 5 | Statistical hypotheses | 6 |
| 6 | Determination of sample size | 6 |
| 7 | General statistical considerations | 6 |
| 7.1 | Analysis populations | <del>6</del> |
| 7.2 | Statistical issues | 7 |
| 7.2.1 | Significance level and confidence intervals | 7 |
| 7.2.2 | Handling of dropouts or missing data | 7 |
| 7.2.3 | Handling of baseline values | 7 |
| 7.2.4 | Interim analyses and data monitoring | 8 |
| 7.2.5 | Multicentre studies | 8 |
| 7.2.6 | Multiplicity | 8 |
| 7.2.7 | Examination of subgroups | 8 |
| 7.2.8 | Checking model assumptions | 8 |
| 7.2.9 | Transformations | 8 |
| 7.2.10 | Handling of outliers and sensitivity analyses | 8 |
| 7.2.11 | Methods for handling multiple time points | 8 |
| 7.2.12 | Descriptive statistics | 8 |
| 8 | Statistical analyses to be used in this study | 9 |
| 8.1 | Disposition of subjects | 9 |
| 8.2 | Demographic and other baseline characteristics | 9 |
| 8.3 | Extent of exposure and measurements of treatment compliance | 9 |
| 8.4 | Analysis of pharmacokinetic variables | 9 |
| 8.4.1 | Primary PK parameter | 10 |
| 8.4.2 | Secondary PK parameters | 11 |
| 8.4.3 | Additional variables | 11 |
| 8.5 | Evaluation and analysis of safety and tolerability | 11 |
| 8.5.1 | Adverse events | 12 |

| 8.5.2 | Laboratory safety variables | 12 |
|---|---|---|
| 8.5.3 | Vitals signs, physical findings, and other observations related to safety | 12 |
| 8.6 | Additional analyses | 12 |
| 8.7 | Changes in the statistical plans from those presented in the clinical study protocol | 12 |
| 8.8 | Execution of statistical analyses | 12 |
| 8.9 | Software | 12 |
| 9 | Reference list | 13 |
| 10 | Appendices | 13 |
| 10.1 | List of tables, figures and graphs | 13 |
| 10.2 | List of subject data listings | 17 |
| 10.3 | Table templates | 19 |

#### 1 Abbreviations

AE Adverse event

AUC Area under the concentration-time curve

BMI Body mass index

BP Blood pressure

C<sub>max</sub> Peak concentration in plasma

C<sub>min</sub> Minimum observed concentration

CV Coefficient of variation

ECG Electrocardiogram

HR Heart rate

IR Immediate release

ITT Intention-to-treat

MR Modified release

PD Parkinson's disease

PG Pharmacogenomic(s)

PK Pharmacokinetic(s)

PP Per-protocol

SAE Serious adverse event

t<sub>1/2</sub> Terminal elimination half-life

t<sub>max</sub> Time to reach peak concentration in plasma

#### 2 General remarks

The purpose of this document is to describe the statistical methodology for this clinical study, including also plans of populations to be used and the plans how the results will be presented.

## 3 Overall study design and plan

This is a phase I, open, repeated dose, randomised PK study in healthy males. The study will be conducted at one centre.

The study will consist of 4 parallel groups (Groups 1-4). All groups will have a crossover design with 4 treatment periods, each lasting for 7 days. The total duration of the study will be approximately 10-15 weeks for each study subject.

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 4 / 28

# 4 Study objectives

#### 4.1 Primary objective

The primary objective is to compare PK of levodopa after repeated administration as follows (Groups 1-4):

#### Group 1:

- A1=50 mg of MR levodopa + 12.5 mg of carbidopa
- B1=50 mg of MR levodopa + 65 mg of carbidopa
- C1=50 mg of MR levodopa + 65 mg of carbidopa + 50 mg of ODM-104
- D1=50 mg of MR levodopa + 65 mg of carbidopa + 100 mg of ODM-104

#### Group 2:

- A2=100 mg of MR levodopa + 25 mg of carbidopa
- B2=100 mg of MR levodopa + 65 mg of carbidopa
- C2=100 mg of MR levodopa + 65 mg of carbidopa + 50 mg of ODM-104
- D2=100 mg of MR levodopa + 65 mg of carbidopa + 100 mg of ODM-104

#### Group 3:

- A3=150 mg of MR levodopa + 37.5 mg of carbidopa
- B3=150 mg of MR levodopa + 65 mg of carbidopa
- C3=150 mg of MR levodopa + 65 mg of carbidopa + 50 mg of ODM-104
- D3=150 mg of MR levodopa + 65 mg of carbidopa + 100 mg of ODM-104

#### Group 4:

- A4=100 mg of IR levodopa + 25 mg of carbidopa (Sinemet®)
- B4=100 mg of MR levodopa + 65 mg of carbidopa
- C4=100 mg of MR levodopa + 25 mg of carbidopa + 100 mg of ODM-104
- D4=100 mg of MR levodopa + 65 mg of carbidopa + 100 mg of ODM-104

The primary objective is to compare PK of 3 different strengths of levodopa after repeated administration in combination with carbidopa and ODM-104.

ODM-104 and carbidopa dose effects will be studied with the 3 MR levodopa strengths and compared with the standard levodopa formulation. Primary comparisons for each of the 4 treatment groups will be performed for levodopa PK between the treatments. The resulting PK data will be used to select the optimal combination of levodopa, carbidopa and ODM-104 for subsequent clinical studies.

#### 4.2 Secondary objectives

The secondary objectives are to determine the PK properties of 3-OMD, carbidopa and ODM-104 in plasma after repeated administration of the different combinations.

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 5 / 28

# 5 Statistical hypotheses

The primary variable for the evaluation of PK of levodopa is  $AUC_{0-24}$  to describe the total levodopa exposure. Primary comparison will be made within levodopa dose level groups, between crossover treatment arms levodopa / 12.5, 25 or 37.5 mg of carbidopa and levodopa / 65 mg of carbidopa / 100 mg of ODM-104. I.e. comparisons A1 vs. D1, A2 vs. D2, A3 vs. D3, and A4 vs. D4 will be the primary ones.

Other crossover comparisons will be performed and considered as secondary. Parallel group comparisons may be performed. The conclusions on possible differences between treatments will be based on both overall evaluation of levodopa concentration-time profiles and formal statistical analyses of PK parameters.

 $H_0$ :  $AUC_{0-24, levodopa/carbidopa /ODM-104} = AUC_{0-24, levodopa/carbidopa}$  $H_1$ :  $AUC_{0-24, levodopa/carbidopa /ODM-104} \neq AUC_{0-24, levodopa/carbidopa}$ 

## 6 Determination of sample size

The sample size estimation is based on earlier ODM-104 phase I study 3112003. Sample size is estimated using the AUC<sub>0-24</sub>. Sample size estimation is based on the results from 12 subjects that completed treatment periods with levodopa 100 mg / carbidopa 25 mg / entacapone 200 mg and MR levodopa 100 mg / carbidopa 65 mg / ODM-104 100 mg. The latter treatment arm with ODM-104 and 65 mg of carbidopa increased exposure by 22% (AUC<sub>0-24</sub> 14022.2 vs. 17092.6). Within subject variability is estimated to be 0.1386 ( $\sqrt{MSE}$  in logarithmic scale). It is assumed that MR levodopa 100 mg / carbidopa 65 mg / ODM-104 100 mg will increase exposure by 40% compared to MR levodopa 100 mg / carbidopa 25 mg.

When the sample size in each sequence is 3 (with a total sample size of 12), a crossover design will have 80% power to detect a difference in means of 0.336 assuming that the within subject variation is 0.139 using a crossover ANOVA with a 0.1 two-sided significance level. To allow drop outs 14 subjects per group and 56 subjects in total will be randomized into this study with 4-treatment, 4-period William's crossover design. This will provide adequate power for the primary comparison. In case there are premature discontinuations the sponsor will decide case-by-case whether replacement subjects will be entered into the study. Replacement subjects will be randomized to go through all 4 treatment periods. Discontinued study subjects are not allowed to re-enter the study.

#### 7 General statistical considerations

#### 7.1 Analysis populations

The datasets derived from individual study subjects will be classified into following three classes prior to database lock and before carrying out any statistical analyses:

• Modified intention-to-treat (mITT) population: all randomized subjects who have received at least one dose of study treatment. The difference between ITT and mITT is that subjects in mITT will be included to have the treatment actually administered. In ITT, subjects are included in the treatment they were intended to be administered.

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 6 / 28

- Per-protocol (PP) population: Subjects who have completed the study according to the protocol without major protocol violations.
- Dosing intervals, where subject experience emesis during the treatment period at Day 7 and following dosing intervals during the period, will be removed from analysis using PP population.
- Periods with PK parameters covering entire Day 7 (e.g. AUC∞) will be excluded from the PP population analysis entirely, in case of emesis.
- If the emesis is experienced at time point 14 hours or thereafter during the last dosing interval, the dosing interval and period will be included into the PP population
- Safety population is the same as the modified ITT population.

The role of each population is described in Table 1.

Table 1. Populations that will be used in tabulations and statistical analyses.

| Primary efficacy | Secondary efficacy | Demographics | Safety variables |
|---|---|---|---|
| variable | variables | Additional variables | |
| PP | PP | mITT | Safety population |
| mITT | mITT | | |

#### 7.2 Statistical issues

#### 7.2.1 Significance level and confidence intervals

90% confidence intervals and p-values will be produced between different treatments. A two-sided significance level of 10% will be considered the level of statistical significance. Confidence intervals and p-values will be presented up to four decimal places.

#### 7.2.2 Handling of dropouts or missing data

In general, missing data or partial data will not be imputed, and statistical analyses will be performed for observed cases only. Possible missing data will be included in statistical calculations via mixed models theory, where missing data can be utilized by setting the subject as random effect in the statistical model. Possible sensitivity analyses may be carried out to evaluate the robustness of the statistical results, that is, particularly the impact of potential outliers.

#### 7.2.3 Handling of baseline values

Screening visit will be used as a baseline for all post baseline variables. If multiple values of a variable are recorded at screening:

- For safety laboratory measurements the last of these values will be used as baseline.
- For ECG the average of these values will be calculated and used as baseline.

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 7/28

#### 7.2.4 Interim analyses and data monitoring

Interim analyses are not planned.

#### 7.2.5 Multicentre studies

This is a single centre study.

#### 7.2.6 Multiplicity

For the primary comparisons, there is only one primary comparison in each group, thus multiplicity correction is not needed. For secondary comparisons, where several treatments are included, all pairwise comparisons will be adjusted according to Tukey method.

#### 7.2.7 Examination of subgroups

No subgroup analyses are planned.

#### 7.2.8 Checking model assumptions

Assumptions for parametric testing will be checked by visual inspection of residuals. If the residuals do not follow normal distribution closely enough, non-parametric comparison methods (e.g. Kruskall-Wallis test for PK variables) or use of transformation will be considered.

#### 7.2.9 Transformations

PK parameters (at least AUC and Cmax) will be analysed after logarithm transformation.

#### 7.2.10 Handling of outliers and sensitivity analyses

If outliers are detected based on residual examination, a sensitivity analysis without the outliers may be performed to evaluate potential impact to the results.

#### 7.2.11 Methods for handling multiple time points

PK parameters C<sub>max</sub>, AUC, t<sub>max</sub> and t<sub>½</sub> will be calculated and used in statistical comparisons. When modelling PK parameters that are calculated by dosing intervals, treatment by dosing interval interaction will be included in the statistical models.

#### 7.2.12 Descriptive statistics

The following statistics will be provided for continuous variables: N, mean, SD, min, median and max. In PK variables also geometric mean and coefficient of variation (CV%) will be calculated. Because log-normal distribution, the formula  $CV\% = 100 \times \sqrt{\exp(\sigma^2 - 1)}$ , where  $\sigma^2$  is MSE of the statistical analysis of log transformed data, will be used. For categorical variables frequency counts and percentages will be presented. All mean, median, standard deviation, and if feasible quartile values will be presented to one more decimal place than the raw values. Minimum and maximum will be presented to the same precision as the raw values.

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 8 / 28

All percentages will be rounded to one decimal place, with the exception of 0 and 100, which will be presented as integers.

## 8 Statistical analyses to be used in this study

#### 8.1 Disposition of subjects

The number of subjects will be tabulated for the following populations:

- Screened
- Randomised
- Modified ITT
- PP
- Safety
- Discontinued study
- Completed study

The disposition and number and reasons for withdrawal and discontinuations will be listed and, if needed, tabulated by treatment sequence. Reasons for excluding subjects or subject periods from pharmacokinetic analyses will be listed. Data from subjects who failed at screening will be included only in the disposition tabulations and data listings.

#### 8.2 Demographic and other baseline characteristics

Demographic and other baseline characteristics will be tabulated by treatment sequence. Medications taken by the subjects before, during, and after the study will be classified by ATC Level 3 and drug name, and will be tabulated and/or listed as appropriate. WHO – DD will be used for coding prior and concomitant medications. No statistical tests will be performed.

#### 8.3 Extent of exposure and measurements of treatment compliance

Each study subject will receive the study treatments under observation of the site personnel. The exposure will be verified by measurement of drug concentrations. Any deviation from the planned compliance and exposure will be listed. Drug administration and plasma concentration data will be listed and tabulated by treatment. The number of subjects exposed to study treatments and the number of doses administered will be tabulated by treatments.

#### 8.4 Analysis of pharmacokinetic variables

Table 2 lists the PK parameters which will be derived from the concentration-time data of levodopa, carbidopa, 3-OMD and, ODM-104.

Table 2. PK parameters to be calculated for levodopa, carbidopa, 3-OMD and ODM-104.

| Parameter | Levodopa | Carbidopa | 3-OMD | ODM-104 |
|----------------------|----------|-----------|-------|------------------|
| $C_{max}$ | $X^1$ | $X^1$ | $X^1$ | $\mathbf{X}^{1}$ |
| $C_{\text{max,tau}}$ | $X^1$ | | | X |

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 9 / 28

| $t_{max}$ | X | X | X | X |
|---|---|---|---|---|
| $t_{max,tau}$ | X | | | X |
| $C_{\min,tau}$ | $X^1$ | | | X |
| C <sub>min,tau,actual</sub> | $X^1$ | | | |
| $AUC_{tau}$ | $X^1$ | | | X |
| $AUC_{0-16}$ | $X^1$ | | | |
| $AUC_{0-24}$ | $X^1$ | $X^1$ | $X^1$ | $\mathbf{X}^{1}$ |
| $\mathrm{AUC}_{\infty}$ | X | | | X |
| $t_{1/2}$ | X | | | X |
| $\lambda_{ m z}$ | X | | | X |
| $C_{\text{max}}/C_{\text{min,tau}}$ | $X^1$ | | | |
| C <sub>max</sub> /C <sub>min,tau,actual</sub> | $X^1$ | | | |
| $C_{\text{max}}/C(16h)$ | $X^1$ | | | |
| PTF <sub>tau</sub> | $X^1$ | | | |
| PTF <sub>0-16h</sub> | $X^1$ | | | |

<sup>1</sup> Statistical analysis will be performed

#### 8.4.1 Primary PK parameter

The primary PK variable for the evaluation of PK of levodopa is AUC0-24 to describe the total levodopa exposure. The primary PK variable will be summarised using descriptive statistics by treatment and analysed using a mixed linear model with 90% CI applicable for the crossover design. The statistical model will include treatment and period as fixed effects and subject as a random effect. Sensitivity analysis adjusted for subject weight and age will be performed.

The following SAS-code for the primary comparison will be applied:

```
proc mixed data=pkparam2 plots=all alpha=0.10;
  class subject trtpcd visit;
  model log_auc = trtpcd visit / ddfm=KR outp=Resid solution;
  random subject;
  lsmeans trtpcd / diff cl alpha=0.10;
  ods output tests3=testCross lsmeans=lsmeansCross
  diffs=diffscross;
  by group;
  run;
```

The following SAS-code for the sensitivity analysis will be applied:

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 10 / 28

```
proc mixed data=pkparam2 plots=all alpha=0.10;
  class subject trtpcd visit;
  model log_auc = trtpcd visit weightkg age / ddfm=KR outp=Resid
  solution;
  random subject;
  lsmeans trtpcd / diff cl alpha=0.10 adjust=tukey ADJDFE=ROW;
  ods output tests3=testCross2 lsmeans=lsmeansCross2
  diffs=diffscross2;
  by group;
  run;
```

#### 8.4.2 Secondary PK parameters

The secondary PK variable is  $C_{min,tau}$ , which is used to describe minimum concentration during the dosing intervals. Statistical evaluation for secondary PK variable will be done using similar methods as for primary variable, except the statistical model will include also the dosing interval as fixed effect.

The following SAS-code for the analysis will be applied:

```
proc mixed data=pkparam2 alpha=0.10;
  class subject trtpcd interval visit;
  model log_auc = trtpcd interval trtpcd*interval visit /
  ddfm=KR outp=Resid solution;
  random subject*visit;
  lsmeans trtpcd trtpcd*interval / diff cl alpha=0.10
  adjust=tukey ADJDFE=ROW;
  ods output tests3=testCross lsmeans=lsmeansCross
  diffs=diffscross;
  by group;
  run;
```

#### 8.4.3 Additional variables

The ratio of the maximum observed concentration (Cmax) in a dosing interval and the observed concentration at the end of the dosing interval, Cmax/Cmin,tau, which is used to describe levodopa fluctuation during the dosing intervals and other PK variables of levodopa, 3-OMD, carbidopa and ODM-104 will be evaluated as additional variables.

Levodopa fluctuation ratios ( $C_{max}/C_{min,tau}$ ,  $C_{max}/C_{(16 h)}$ , PTF<sub>tau</sub> and PTF<sub>(0-16)</sub>, and AUC<sub>0-24</sub>,  $C_{max}$  and  $C_{min,tau}$  will be the main PK variables of interest.

Drug concentrations will be tabulated by time and treatment with descriptive statistics.

#### 8.5 Evaluation and analysis of safety and tolerability

Safety will be evaluated by recording heart rate, systolic and diastolic blood pressure, 12-lead electrocardiogram (ECG), physical examination findings, laboratory safety assessments and

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 11 / 28

adverse events (AEs). Suicidality will be assessed with the Columbia-Suicide Severity Rating Scale (C-SSRS).

#### 8.5.1 Adverse events

Adverse events (AEs) reported after administration of the study treatment will be classified by System organ classes (SOC) and preferred terms using the MedDRA dictionary.

The number and proportion (%) of subjects having each AE will be given by treatment group. The numbers will be additionally broken down by severity (mild, moderate, severe) and by the causality (related, not related).

All serious adverse events (SAEs) and other significant AEs will be evaluated case by case. Additionally, narrative descriptions will be included in the study report for all SAEs and certain other significant AEs.

#### 8.5.2 Laboratory safety variables

Laboratory values and changes from baseline (screening value) in laboratory values will be summarised using descriptive statistics. The number and proportion of subjects with laboratory values outside the normal range will be summarised by visit for each laboratory analyte. Unscheduled laboratory measurements will not be used in tables. They will be included in the listings.

#### 8.5.3 Vitals signs, physical findings, and other observations related to safety

Vital signs (systolic and diastolic BP and HR) at each visit and change from baseline (screening value) in each vital sign will be summarised using descriptive statistics. 12-lead ECG parameters at each time point and change from baseline (screening value) will be summarised using descriptive statistics. Physical examination and C-SSRS findings will be tabulated.

#### 8.6 Additional analyses

# 8.7 Changes in the statistical plans from those presented in the clinical study protocol

#### 8.8 Execution of statistical analyses

Statistical analyses will be performed by or under the supervision of the Department of Biostatistics and Support Functions of Orion Pharma.

#### 8.9 Software

Statistical analyses, tables and subject data listings will be performed with SAS® for Windows version 9.4 (SAS Institute Inc., Cary, NC, USA).

DNO 090017ff81c5a601 / 1.0 Confidential Approved 12 / 28

# 9 Reference list

1. SAS, Institute Inc., Cary, NC, USA.

# 10 Appendices

# 10.1 List of tables, figures and graphs

# 14 Post-text tables and figures

# 14.1 Demographic data

| Table 14.1.1 | Disposition of subjects |
|---|---|
| Table 14.1.2.1 | Reasons for excluding data from the statistical analyses of pharmacokinetic parameters |
| Table 14.1.2.2 | Reasons for study discontinuation |
| Table 14.1.3 | Demographic and other baseline characteristics |
| Table 14.1.4 | Medical history and current medical conditions |
| Table 14.1.5.1 | Prior treatments |
| Table 14.1.5.2 | Concomitant treatments during study treatment periods |
| Table 14.1.5.3 | Concomitant treatments after end of study treatment |
| Table 14.1.6 | Extent of exposure |

#### 14.2 Pharmacokinetic data

| Table 14.2.1.1 | Levodopa concentration (ng/ml) |
|---|---|
| Table 14.2.1.2.1 | AUCtau (h*ng/mL) of levodopa |
| Table 14.2.1.2.2 | Statistical analysis for AUCtau of levodopa |
| Table 14.2.1.3.1 | AUC0-24 (h*ng/mL) of levodopa |
| Table 14.2.1.3.2 | Statistical analysis for AUC0-24 of levodopa |
| Table 14.2.1.4.1 | AUC0-16 (h*ng/mL) of levodopa |
| Table 14.2.1.4.2 | Statistical analysis for AUC0-16 of levodopa |
| Table 14.2.1.5 | AUCinf (h*ng/mL) of levodopa |
| Table 14.2.1.6.1 | Cmax,tau (ng/mL) of levodopa |
| Table 14.2.1.6.2 | Statistical analysis for Cmax,tau of levodopa |
| Table 14.2.1.7.1 | Cmax (ng/ml) of levodopa |
| Table 14.2.1.7.2 | Statistical analysis for Cmax of levodopa |
| Table 14.2.1.8.1 | Cmin,tau (ng/mL) of levodopa |
| Table 14.2.1.8.2 | Statistical analysis for Cmin,tau (ng/mL) of levodopa |
| Table 14.2.1.8.3 | Actual Cmin,tau (ng/mL) of levodopa |
| Table 14.2.1.8.4 | Statistical analysis for actual Cmin,tau (ng/mL) of levodopa |
| Table 14.2.1.9.1 | Cmax / Cmin ratio tau of levodopa |
| Table 14.2.1.9.2 | Statistical analysis of Cmax / Cmin ratio tau of levodopa |

DNO 090017ff81c5a601 / 1.0 Confidential Approved 13 / 28

| 1 | <del>-</del> |
|---|---|
| Table 14.2.1.9.3 | Actual Cmax / Cmin ratio tau of levodopa |
| Table 14.2.1.9.4 | Statistical analysis of actual Cmax / Cmin ratio tau of levodopa |
| Table 14.2.1.10.1 | Cmax / C(16h) of levodopa |
| Table 14.2.1.10.2 | Statistical analysis of Cmax / C(16h) of levodopa |
| Table 14.2.1.11 | tmax,tau (h) of levodopa |
| Table 14.2.1.12 | tmax (h) of levodopa |
| Table 14.2.1.13 | t1/2 (h) of levodopa |
| Table 14.2.1.14 | Lambda z of levodopa |
| Table 14.2.1.15.1 | PTFtau of levodopa |
| Table 14.2.1.15.2 | Statistical analysis for PTFtau of levodopa |
| Table 14.2.1.16.1 | PTF0-16 of levodopa |
| Table 14.2.1.16.2 | Statistical analysis for PTF0-16 of levodopa |
| Table 14.2.2.1 | Carbidopa concentrations (ng/ml) |
| Table 14.2.2.2.1 | AUC0-24 (h*ng/mL) of Carbidopa |
| Table 14.2.2.2.2 | Statistical analysis for AUC0-24 (h*ng/mL) of Carbidopa |
| Table 14.2.2.3.1 | Cmax (ng/ml) of Carbidopa |
| Table 14.2.2.3.2 | Statistical analysis for Cmax (ng/ml) of Carbidopa |
| Table 14.2.2.4 | tmax (h) of Carbidopa |
| Table 14.2.3.1 | 3-ODM concentrations (ng/ml) |
| Table 14.2.3.2.1 | AUC0-24 (h*ng/mL) of 3-ODM |
| Table 14.2.3.2.2 | Statistical analysis for AUC0-24 (h*ng/mL) of 3-ODM |
| Table 14.2.3.3.1 | Cmax (ng/ml) of 3-ODM |
| Table 14.2.3.3.2 | Statistical analysis for Cmax (ng/ml) of 3-ODM |
| Table 14.2.3.4 | tmax (h) of 3-ODM |
| Table 14.2.4.1 | ODM-104 concentrations (ng/ml) |
| Table 14.2.4.2 | AUC0tau (h*ng/mL) of ODM-104 |
| Table 14.2.4.3 | AUC0-24 (h*ng/mL) of ODM-104 |
| Table 14.2.4.4 | Statistical analysis of AUC0-24 (h*ng/mL) of ODM-104 |
| Table 14.2.4.5 | AUCinf (h*ng/mL) of ODM-104 |
| Table 14.2.4.6 | Cmax,tau (ng/ml) of ODM-104 |
| Table 14.2.4.7 | Cmax (ng/ml) of ODM-104 |
| Table 14.2.4.8 | Statistical analysis of Cmax (ng/ml) of ODM-104 |
| Table 14.2.4.9 | Cmin,tau (ng/ml) of ODM-104 |
| Table 14.2.4.10 | tmax,tau (h) of ODM-104 |
| Table 14.2.4.11 | tmax (h) of ODM-104 |
| Table 14.2.4.12 | t½ (h) of ODM-104 |
| Table 14.2.4.13 | Lambda z of ODM-104 |
| - | |

# 14.3 Safety data

| Table 14.3.1.1 | Summary of adverse events during study treatment (subject and event count) |
|---|---|
| Table 14.3.1.2 | Adverse events during study treatment (subject and event count) |

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 14 / 28

| T 11 14212 | |
|---|---|
| Table 14.3.1.3 | Adverse events during study treatment by severity (subject count) |
| Table 14.3.1.4 | Adverse events related to study treatment (subject and event count) |
| Table 14.3.1.5 | Adverse events during study treatment by severity and causality (event count) |
| Table 14.3.1.6 | Adverse events before start of study treatment (subject and event count) |
| Table 14.3.1.7 | Adverse events at the end of study (subject and event count) |
| Table 14.3.2.1 | Summary listing of deaths, other serious and significant adverse events |
| Table 14.3.2.2 | Listing of deaths |
| Table 14.3.2.3 | Listing of serious adverse events |
| Table 14.3.2.4 | Listing of adverse events leading to premature discontinuation |
| Table 14.3.2.5 | Listing of other significant adverse events |
| Table 14.3.2.6 | Listing of special situations |
| Table 14.3.3.1 | Summary listing of narratives of deaths, other serious and significant adverse events |
| Table 14.3.4 | Listing of significant abnormal laboratory values |
| Table 14.3.5.1.1 | Haematology |
| Table 14.3.5.1.2 | Changes from baseline in haematology |
| Table 14.3.5.1.3 | Shift tables for haematology variables |
| Table 14.3.5.2.1 | Chemistry |
| Table 14.3.5.2.2 | Changes from baseline in chemistry |
| Table 14.3.5.2.3 | Shift tables for chemistry variables |
| Table 14.3.5.3 | Serology |
| Table 14.3.5.4.1 | Urinalysis |
| Table 14.3.5.4.2 | Shift tables for urinalysis variables - Safety population |
| Table 14.3.6.1.1 | Supine heart rate (bpm) |
| Table 14.3.6.1.2 | Changes from baseline in supine heart rate (bpm) |
| Table 14.3.6.2.1 | Supine diastolic blood pressure (mmHg) |
| Table 14.3.6.2.2 | Changes from baseline in supine diastolic blood pressure (mmHg) |
| Table 14.3.6.3.1 | Supine systolic blood pressure (mmHg) |
| Table 14.3.6.3.2 | Changes from baseline in supine systolic blood pressure (mmHg) |
| Table 14.3.7.1.1 | Summary of 12-lead ECG findings |
| Table 14.3.7.1.2 | Shift table for 12-lead ECG findings |
| Table 14.3.7.2.1 | PR interval (ms) |
| Table 14.3.7.2.2 | Changes from baseline in PR interval (ms) |
| Table 14.3.7.3.1 | QRS interval (ms) |
| Table 14.3.7.3.2 | Changes from baseline in QRS interval (ms) |
| Table 14.3.7.4.1 | RR interval (ms) |
| Table 14.3.7.4.2 | Changes from baseline in RR interval (ms) |
| Table 14.3.7.5.1 | QT interval (ms) |
| Table 14.3.7.5.2 | Changes from baseline in QT interval (ms) |
| | 3 |
| Table 14.3.7.7.1 | QTc [Fridericia] interval (ms) |
| Table 14.3.7.7.2 | Changes from baseline in QTc [Fridericia] interval (ms) |
| 14010 17.3.7.7.2 | Changes from oaseine in Q1e [1 factions] interval (ins) |

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 15 / 28

| Table 14.3.7.8.1 | QT interval (categorical analyses) |
|---|---|
| Table 14.3.7.8.2 | Changes from baseline in QT interval (categorical analyses) |
| Table 14.3.7.10.1 | QTc [Fridericia] interval (categorical analyses) |
| Table 14.3.7.10.2 | Changes from baseline in QTc [Fridericia] interval (categorical analyses) |
| Table 14.3.1.8 | Physical examination |
| Table 14.3.1.9 | Suicidality assessment by C-SSRS during treatment |
| Table 14.3.1.9.1 | Suicidality assessment by C-SSRS - Screening |

# 14.4 Figures

| Figure 14.4.1.1 | Mean $\pm$ (SEM) levodopa concentration profile |
|------------------|----------------------------------------------------------|
| Figure 14.4.1.2 | Individual levodopa concentration profiles |
| Figure 14.4.1.3 | Individual levodopa concentration profiles by subject |
| Figure 14.4.2.1 | Mean $\pm$ (SEM) carbidopa concentration profile |
| Figure 14.4.2.2 | Individual carbidopa concentration profiles |
| Figure 14.4.2.3 | Individual carbidopa concentration profiles by subject |
| Figure 14.4.3.1 | Mean $\pm$ (SEM) 3-OMD concentration profile |
| Figure 14.4.3.2 | Individual 3-OMD concentration profiles |
| Figure 14.4.3.3 | Individual 3-OMD concentration profiles by subject |
| Figure 14.4.4.1 | Mean ± (SEM) ODM-104 concentration profile |
| Figure 14.4.4.2 | Individual ODM-104 concentration profiles |
| Figure 14.4.4.3 | Individual ODM-104 concentration profiles by subject |
| Figure 14.4.5.1 | Mean ± (SEM) heart rate - Supine |
| Figure 14.4.5.2 | Mean ± (SEM) change of heart rate - Supine |
| Figure 14.4.5.3 | Individual profiles of heart rate - Supine |
| Figure 14.4.6.1 | Mean ± (SEM) systolic blood pressure - Supine |
| Figure 14.4.6.2 | Mean ± (SEM) change of systolic blood pressure - Supine |
| Figure 14.4.6.3 | Individual profiles of systolic blood pressure - Supine |
| Figure 14.4.7.1 | Mean ± (SEM) diastolic blood pressure - Supine |
| Figure 14.4.7.2 | Mean ± (SEM) change of diastolic blood pressure - Supine |
| Figure 14.4.7.3 | Individual profiles of diastolic blood pressure - Supine |
| Figure 14.4.8.1 | Mean $\pm$ (SEM) of PR interval |
| Figure 14.4.8.2 | Mean ± (SEM) change of PR interval |
| Figure 14.4.8.3 | Individual profiles of PR interval |
| Figure 14.4.9.1 | Mean ± (SEM) of QRS interval |
| Figure 14.4.9.2 | Mean ± (SEM) change of QRS interval |
| Figure 14.4.9.3 | Individual profiles of QRS interval |
| Figure 14.4.10.1 | Mean $\pm$ (SEM) of RR interval |
| Figure 14.4.10.2 | Mean ± (SEM) change of RR interval |
| Figure 14.4.10.3 | Individual profiles of RR interval |

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 16 / 28

| Figure 14.4.11.1 | Mean $\pm$ (SEM) of QT interval |
|------------------|------------------------------------------|
| Figure 14.4.11.2 | Mean $\pm$ (SEM) change of QT interval |
| Figure 14.4.11.3 | Individual profiles of QT interval |
| Figure 14.4.12.1 | Mean $\pm$ (SEM) of QTcB interval |
| Figure 14.4.12.2 | Mean $\pm$ (SEM) change of QTcB interval |
| Figure 14.4.12.3 | Individual profiles of QTcB interval |
| Figure 14.4.13.1 | Mean $\pm$ (SEM) of QTcF interval |
| Figure 14.4.13.2 | Mean $\pm$ (SEM) change of OTcF interval |
| Figure 14.4.13.3 | Individual profiles of QTcF interval |

## 10.2 List of subject data listings

#### 16.2. SUBJECT DATA LISTINGS

The section headings are given in italics, and other headings are actual listings for data.

- 16.2.1 Discontinued subjects and disposition
- 16.2.1.1 Study discontinuations
- 16.2.1.2 Disposition of subjects
- 16.2.1.3 Study dates
- 16.2.2 Protocol deviations
- 16.2.2.1 Protocol deviations
- 16.2.3 Subjects and observations excluded from efficacy analyses/statistical analyses of pharmacokinetic parameters
- 16.2.3.1 Reasons for excluding observations from efficacy analyses/PK parameters
- 16.2.4 Demographic data
- 16.2.4.1 Demographic and other baseline characteristics
- 16.2.4.2 Medical history and current medical conditions
- 16.2.4.3 Concomitant treatments
- 16.2.5 Compliance data and/or drug concentration data
- 16.2.5.1 Concentration data of ODM-104
- 16.2.5.2 Concentration data of levodopa carbidopa and 3-OMD
- 16.2.6 Pharmacokinetic data
- 16.2.6.1 Study treatment administration and blood sampling times

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 17 / 28

| 16.2.6.2 | Pharmacokinetic parameters of ODM-104 |
|---|---|
| 16.2.6.3 | Pharmacokinetic parameters of levodopa |
| 16.2.6.4 | Pharmacokinetic parameters of carbidopa |
| 16.2.6.5 | Pharmacokinetic parameters of 3-OMD |
| 16.2.7 Advers | e events |
| 16.2.7.1 | Adverse events before start of study treatment |
| 16.2.7.2 | Adverse events after start of study treatment |
| 16.2.8 Labora | atory measurements |
| 16.2.8.1 | Laboratory measurements |
| 16.2.9 Vital si | igns, physical findings and other observations related to safety |
| 16.2.9.1 | Vital signs |
| 16.2.9.2 | Physical examination |
| 16.2.9.3 | 12-lead ECG |
| 16.2.9.4 | Suicidality assessments using C-SSRS |
| 16.2.10.1 | Water intake and meals |

Note! In case no observation fulfils the listing criteria's, e.g. no discontinuations, an empty list is produced.

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 18 / 28

### 10.3 Table templates

Examples of tables.

STUDY 3112005

DRAFT

Page: 1 (1)

Table 14.1.1 Disposition of subjects Modified Intention to treat population

| | Group 1<br>(N=XX) | Group 2<br>(N=XX) | Group 3<br>(N=XX) | Group 4<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|---|---|
| | n (%) | n (%) | n (%) | n (%) | n (%) |
| Screened | | | | | 82 |
| Randomised | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) |
| Intent-to-treat population | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) |
| Per-protocol population | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) |
| Safety population | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) |
| Completed study | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| Discontinued study | X (XX.X) | X ( X.X) | X (XX.X) | X ( X.X) | X (XX.X) |

Program: T\_14\_1\_1\_Disposition of subjects.sas Date: 23MAY17:08:17

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 19 / 28

DRAFT

Page: 1 (2)

Table 14.1.3 Demographic and other baseline characteristics Modified Intention to treat population

| | | Group 1 (N=XX) | Group 2<br>(N=XX) | Group 3 (N=XX) | Group 4<br>(N=XX) | Total<br>(N=XX) |
|---|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) | n (%) |
| Gender<br>Race | MALE<br>CAUCASIAN | XX ( XXX)<br>XX ( XXX) | XX (XXX)<br>XX (XX.X) | XX ( XXX)<br>XX ( XXX) | XX (XXX)<br>XX (XX.X) | XX (XXX)<br>XX (XX.X) |
| | ASIAN | X (X.X) | X ( X.X) | X ( X.X) | X ( X.X) | X ( X.X) |
| Age (years) | N | XX | XX | XX | XX | XX |
| rige (years) | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX | XX | XX |
| Weight (kg) | N | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.X | X.X | XX.X | XX.X | X.X |
| | Min | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Max | XX | XX | XXX | XX | XXX |
| Height (cm) | N | XX | XX | XX | XX | XX |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | X.X | X.X | X.X | X.X | X.X |
| | Min | XXX | XXX | XXX | XXX | XXX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X | XXX.X |
| | Max | XXX | XXX | XXX | XXX | XXX |

Program: T\_14\_1\_3\_Demographics and other baseline characteristics.sas

Date: 23MAY17:08:19

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 20 / 28

Table 14.2.1.2.1 AUCtau (h\*ng/mL) of levodopa Per protocol population

| | | A1<br>(N=XX) | B1<br>(N=XX) | C1<br>(N=XX) | D1<br>(N=XX) |
|---|---|---|---|---|---|
| AUC 0-3.5h | N | XX | XX | XX | XX |
| 1100 0 3:311 | Gmean | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | Mean | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XXXX.X | XXXX.X | XXXX.X | XXX.X |
| | Median | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | Max | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| AUC 3.5-7h | N | XX | XX | XX | XX |
| 1100 3.3 711 | Gmean | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | Mean | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | SD | XXXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | Median | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | Max | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| AUC 7-10.5h | N | XX | XX | XX | XX |
| 1100 / 10:011 | Gmean | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | Mean | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | SD | XXXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | Median | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | Max | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| AUC 10.5-14h | N | XX | XX | XX | XX |
| | Gmean | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | Mean | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | SD | XXX.XX | XXX.XX | XXX.XX | XXX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | Median | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | Max | XXXX.X | XXXX.X | XXXX.X | XXXX.X |

Program: T\_14\_2\_1\_2\_1\_Levodopa AUC\_tau.sas Date: 23MAY17:08:38

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 21 / 28

DRAFT

Page: 1 (4)

Table 14.2.1.3.1 AUC0-24 (h\*ng/mL) of levodopa Per protocol population

| | | A1<br>(N=XX) | B1<br>(N=XX) | C1<br>(N=XX) | D1<br>(N=XX) |
|---|---|---|---|---|---|
| AUC0 24h | N | XX | XX | XX | XX |
| | Gmean | XXXXX.XX | XXXXX.XX | XXXXX.XX | XXXXX.XX |
| | Mean | XXXXX.XX | XXXXX.XX | XXXXX.XX | XXXXX.XX |
| | SD | XXXX.XX | XXXX.XX | XXXX.XX | XXXX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XXXX.X | XXXX.X | XXXX.X | XXXX.X |
| | Median | XXXXX.XX | XXXXX.XX | XXXXX.XX | XXXXX.XX |
| | Max | XXXXX.X | XXXXX.X | XXXXX.X | XXXXX.X |

Program: T\_14\_2\_1\_3\_1\_Levodopa AUC0-24.sas Date: 23MAY17:08:40

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 22 / 28

DRAFT

Page: 1 (8)

Table 14.2.1.3.2 Statistical analysis for AUC0-24 of levodopa Per protocol population

#### Analysis of variance

| | | Estimate | | 90% | |
|---|---|---|---|---|---|
| Effect | | (Geometric Mean) | Stderr | Confidence Interval | P-value |
| Fixed Effects | | | | | |
| Formulation | | | | | X.XXXX |
| Period | | • | | | X.XXXX |
| Least Square Me | eans | | | | |
| Formulation A1 | | XXXXX.XXX | X.XXX | XX(XXXXX.XX,XXXXXXXXXXXXXXXXXXXXXXXXXXX | <.xxxx |
| Formulation B1 | | XXXXX.XXX | | (XXXXXX.XX ,XXXXX.XX) | <.xxxx |
| Formulation C1 | | XXXXX.XXX | X.XXX | (XXXXXX.XX ,XXXXX.XX) | <.xxxx |
| Formulation D1 | | XXXXX.XXX | X.XXX | XX(XXXXX.XX,XXXXXXXXXXXXXXXXXXXXXXXXXXX | <.XXXX |
| Differences in | Least | Square Means | | | |
| Formulation A1 | | X.XXXXXXX | X.XXX | XX( X.XXXX , X.XXXX) | X.XXXX |
| Formulation A1 | . C1 | X.XXXXXX | X.XXX | XX( X.XXXX, X.XXXX) | X.XXXX |
| Formulation A1 | . D1 | X.XXXXX | X.XXX | XX( X.XXXX, X.XXXX) | X.XXXX |
| Formulation B1 | . C1 | X.XXXXX | X.XXX | XX( X.XXXX, X.XXXX) | X.XXXX |
| Formulation B1 | . D1 | X.XXXXXX | X.XXX | XX( X.XXXX , X.XXXX) | X.XXXX |
| Formulation C1 | . D1 | X.XXXXXXX | X.XXX | XX( X.XXXX , X.XXXX) | X.XXXX |

Program: T\_14\_2\_1\_3\_2\_Levodopa statistical analysis for AUC0-24.sas Date: 23MAY17:08:40

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 23 / 28

DRAFT

Page: 1 (5)

Table 14.3.1.1 Summary of adverse events during study treatment (subject and event count) Safety population

| | | | A1<br>(N=XX) | | B1<br>(N=XX) | | C1<br>(N=XX) | | D1<br>(N=XX) |
|---|---|---|---|---|---|---|---|---|---|
| | | | n (%) | | n (%) | | n (%) | | n (%) |
| Subject count | AEs | Х | (XX.X) | Х | (XX.X) | Х | (XX.X) | Х | (XX.X) |
| | Related AEs | X | (XX.X) | X | (XX.X) | Χ | (XX.X) | X | (XX.X) |
| | AEs leading to | | | | | | | | |
| | discontinuation of study | | | | | | | | |
| | Mild AEs | X | (XX.X) | X | (XX.X) | X | (XX.X) | Χ | (XX.X) |
| | Moderate AEs | Х | (XX.X) | Χ | (XX.X) | Х | (XX.X) | Χ | (XX.X) |
| | Severe AEs | | | | | | | | |
| | SAEs | | | | | | | | |
| Event count | AEs | | XX | | XX | | XX | | XX |
| | Related AEs | | X | | XX | | XX | | XX |
| | AEs leading to | | | | | | | | |
| | discontinuation of study | | | | | | | | |
| | Mild AEs | | X | | XX | | X | | XX |
| | Moderate AEs | | X | | X | | XX | | X |
| | Severe AEs | | | | | | | | |
| | SAEs | | | | | | | | |

Program: T\_14\_3\_1\_1\_Summary of AEs.sas Date: 23MAY17:08:57

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 24 / 28

DRAFT

Page: 1 (10)

Table 14.3.1.2 Adverse events during study treatment (subject and event count) Safety population

| - | B1 | C1 | A1 | D1 |
|---|---|---|---|---|
| Contain One of Class | (N=XX) | (N=XX) | (N=XX) | (N=XX) |
| System Organ Class | Subjects Events | Subjects Events | | • |
| Preferred Term | n (%) n | n (%) n | n (%) n | n (%) n |
| Cardiac disorders | | | | |
| Total | X ( X.X) X | X ( X.X) X | | |
| Cardiovascular insufficiency | 21 (21,21) 21 | X ( X.X) X | | |
| Palpitations | X (X.X) X | $\Lambda (\Lambda \cdot \Lambda) \Lambda$ | | |
| Gastrointestinal disorders | | | | |
| Total | X (XX.X) X | X (XX.X) X | X (XX.X) X | |
| Abdominal discomfort | X ( X.X) X | X (X.X) X | | |
| Abdominal pain | | X (X.X) X | | |
| Abdominal pain lower | | | X (X.X) X | |
| Diarrhoea | X (XX.X) X | X (X.X) X | | |
| Flatulence | | X (X.X) X | X (X.X) X | |
| Gingival bleeding | X (X.X) X | | | |
| General disorders and administration site | | | | |
| conditions | | | | |
| Total | | | | X (X.X) X |
| Fatigue | | | | X ( X.X) X |
| Infections and infestations | | | | |
| Total | X ( X.X) X | X (X.X) X | X (X.X) X | X (X.X) X |
| Gingivitis | | | | X (X.X) X |
| Nasopharyngitis | X (X.X) X | X ( X.X) X | X ( X.X) X | |
| Injury, poisoning and procedural complications | | | | |
| Total | X (X.X) X | | X (X.X) X | |
| Muscle strain | X (X.X) X | | | |
| Thermal burn | | | X (X.X) X | |

Program: T\_14\_3\_1\_2\_AEs by SOC and PT.sas Date: 23MAY17:08:58

DRAFT

Page: 1 (24)

Table 14.3.5.1.1 Haematology Safety population

Laboratory variable=B-Erythrocytes - 10E12/l

| | | N | Mean | SD | Minimum | Median | Maximum |
|-----------|-----------|----|-------|-------|---------|--------|---------|
| Treatment | | | | | | | |
| _ | Screening | XX | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| A1 | Period 1 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 2 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 3 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 4 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| B1 | Period 1 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 2 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 3 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 4 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| C1 | Period 1 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 2 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 3 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 4 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| D1 | Period 1 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 2 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 3 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 4 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| A2 | Period 1 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 2 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 3 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |
| | Period 4 | X | X.XXX | X.XXX | X.XX | X.XXX | X.XX |

Program: T\_14\_3\_5\_1\_1\_Haematology.sas Date: 23MAY17:10:58

DRAFT

Page: 1 (16)

Table 14.3.7.2.2 Changes from baseline in PR interval (ms) Safety population

| Treatment | | N | Mean | SD | Minimum | Median | Maximu<br>m |
|---|---|---|---|---|---|---|---|
| _ | Screening | Х | | | | | |
| A1 | Period 1 DAY -1 | X | -x.xx | XX.XX | -xx.x | -X.XX | XX.X |
| 111 | Period 1 DAY 1: 0-2 H BEFORE FIRST DOSE | X | | | | | |
| | Period 1 DAY 6: 1-2 H AFTER 7 H DOSE | X | -x.xx | XX.XX | -xx.x | -X.XX | XX.X |
| | Period 1 DAY 7: 0-2 H BEFORE FIRST DOSE | Х | X.XX | XX.XX | -x.x | X.XX | XX.X |
| | Period 1 DAY 7: 1-2 H AFTER 7 H DOSE | X | X.XX | X.XX | -x.x | -x.xx | XX.X |
| | Period 2 DAY -1 | X | X.XX | X.XX | -X.X | X.XX | X.X |
| | Period 2 DAY 1: 0-2 H BEFORE FIRST DOSE | X | | | | | |
| | Period 2 DAY 6: 1-2 H AFTER 7 H DOSE | X | -X.XX | XX.XX | -XX.X | -X.XX | XX.X |
| | Period 2 DAY 7: 0-2 H BEFORE FIRST DOSE | X | X.XX | X.XX | -X.X | X.XX | XX.X |
| | Period 2 DAY 7: 1-2 H AFTER 7 H DOSE | X | X.XX | X.XX | -X.X | X.XX | XX.X |
| | Period 3 DAY -1 | X | -XX.XX | XX.XX | -XX.X | -XX.XX | -X.X |
| | Period 3 DAY 1: 0-2 H BEFORE FIRST DOSE | X | • | | | • | • |
| | Period 3 DAY 6: 1-2 H AFTER 7 H DOSE | X | -X.XX | X.XX | -XX.X | -X.XX | X.X |
| | Period 3 DAY 7: 0-2 H BEFORE FIRST DOSE | X | -X.XX | X.XX | -XX.X | X.XX | X.X |
| | Period 3 DAY 7: 1-2 H AFTER 7 H DOSE | X | -X.XX | XX.XX | -XX.X | -X.XX | X.X |
| | Period 4 DAY -1 | X | X.XX | XX.XX | -X.X | -X.XX | XX.X |
| | Period 4 DAY 1: 0-2 H BEFORE FIRST DOSE | X | | • | | | |
| | Period 4 DAY 6: 1-2 H AFTER 7 H DOSE | X | X.XX | XX.XX | -XX.X | -X.XX | XX.X |
| | Period 4 DAY 7: 0-2 H BEFORE FIRST DOSE | X | -X.XX | X.XX | -XX.X | X.XX | X.X |
| | Period 4 DAY 7: 1-2 H AFTER 7 H DOSE | X | -X.XX | X.XX | -XX.X | X.XX | X.X |

Screening value is considered as baseline

Program: T\_14\_3\_7\_2\_2\_Change from bl in PR interval.sas

Date: 23MAY17:09:10

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 27 / 28

DRAFT

Page: 1 (4)

Table 14.3.1.9 Suicidality assessment by C-SSRS during treatment Safety population

| | | A1<br>(N=13) | B1<br>(N=14) | C1<br>(N=14) | D1<br>(N=13) |
|---|---|---|---|---|---|
| | | n (%) | n (%) | n (%) | n (%) |
| CSS02-Wish to be Dead | NO | XX ( XXX) | XX ( XXX) | XX ( XXX) | XX ( XXX) |
| CSS02-Non-Specific Suicidal Thought | NO | XX (XXX) | XX (XXX) | XX (XXX) | XX ( XXX) |
| CSS02-Actual Attempt | NO | XX (XXX) | XX ( XXX) | XX (XXX) | XX ( XXX) |
| CSS02-Non-suicidal Self-injurious Behav | NO | XX (XXX) | XX ( XXX) | XX (XXX) | XX ( XXX) |
| CSS02-Interrupted Attempt | NO | XX (XXX) | XX ( XXX) | XX (XXX) | XX ( XXX) |
| | NA | X ( X.X) | X (X.X) | X ( X.X) | X ( X.X) |
| CSS02-Aborted Attempt | NO | XX ( XXX) | XX ( XXX) | XX (XXX) | XX ( XXX) |
| CSS02-Preparatory Acts/Behavior | NO | XX (XXX) | XX ( XXX) | XX (XXX) | XX ( XXX) |
| | NA | X ( X.X) | X (X.X) | X ( X.X) | X ( X.X) |
| CSS02-Suicidal Behavior | NO | XX (XXX) | XX (XXX) | XX (XXX) | XX ( XXX) |
| CSS02-Suicide | NO | XX ( XXX) | XX (XXX) | XX (XXX) | XX ( XXX) |

Program: T\_14\_3\_9\_C-SSRS.sas Date: 23MAY17:09:14

DNO 090017ff81c5a601 / 1.0 Confidential **Approved** 28 / 28



# 3112005 Statistical Analysis Plan

# Written by: Vahteristo Mikko

| Date dd.mm.yyyy (UTC) | Justification | Electronically signed by |
|-----------------------|---------------|---------------------------|
| 13.06.2017 07:21:31 | Approved | Vahteristo Mikko (mikvah) |
| 13.06.2017 07:46:02 | Approved | Ellmen Juha (juhael) |
| 14.06.2017 04:37:59 | Approved | Holopainen Aila (ailaho) |

DNO 090017ff81c5a601 / 1.0 Confidential Approved